CLINICAL TRIAL: NCT05533736
Title: Feasibility and Usability of Mobile Applications for Monitoring Cutaneous Leishmaniasis Treatment in Colombia: 2019-2021
Brief Title: Feasibility and Usability of Mobile Applications for Monitoring Cutaneous Leishmaniasis Treatment in Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Internacional de Entrenamiento e Investigaciones Médicas (Other)
Collaborators: Universidad Icesi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 201875
Record Dates: First submitted 2022-09-01; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Cutaneous Leishmaniasis, American
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community based strategy to follow-up pactientes with Cutaneous Leishmaniasis (Experimental): Patients with cutaneous leishmaniasis are followed with the Guaral+ST app by Community Health Leaders. This intervention was not randomized
  Interventions: Other: Community based strategy to follow-up pactientes with Cutaneous Leishmaniasis
- Control group: Standard of care (No Intervention): Control group: Standard of Care: Registers historical patients with cutaneous leishmaniasis is followed in the health facility by physicians according to national guidelines.

INTERVENTIONS:
Other: Community based strategy to follow-up pactientes with Cutaneous Leishmaniasis — Community Health leaders follow patients using the Guaral+ST app at final of treatment, and on days 90 and 180 after initiating the treatment.
  Arms: Community based strategy to follow-up pactientes with Cutaneous Leishmaniasis

SUMMARY:
An effectiveness-implementation sequential explanatory hybrid design type 2 was performed in two rural communities of Colombia. A quasi-experimental study with historical control (standard of care) was designed to estimate the effectiveness of community-based intervention using the Guaral+ST mobile application (app). Three implementation outcomes were evaluated: acceptability and usability by qualitative methods, and fidelity by quantitative methods

DETAILED DESCRIPTION:
An effectiveness-implementation sequential explanatory hybrid design type 2 using mixed methods was performed in 2020 and 2021 in two study sites: Pueblo Rico, Risaralda, and Rovira, Tolima. A quasi-experimental study with historical control (standard of care) was designed to evaluate the effectiveness of the community-based intervention supported by mHealth, in terms of monitoring of treatment of patients with cutaneous leishmaniasis. The effectiveness indicators i. number of follow-up contacts, ii. Adherence to treatment, iii. adverse drug reactions, and iv. the therapeutic response were compared between the intervention and control groups.

After the effectiveness evaluation was completed, three outcomes were assessed to inform the implementation of the community-based use of the app: acceptability, usability, and fidelity.

ELIGIBILITY:
Inclusion Criteria:

Patients followed by CHL with the app (effectiveness evaluation):

* Diagnosis confirmed by microscopy of tissue smear or culture
* Any age and gender
* Medical prescription for antileishmanial treatment
* Approved and signed informed consent
* Availability of CHL to monitor treatment of the patients in the community

Inclusion Criteria patients who received the standard of care (effectiveness evaluation):

* Clinical records of patients with confirmed CL at most two years prior to the start of this study
* Any age and gender
* Received antileishmanial treatment based on national guidelines

Inclusion criteria for participants of implementation evaluation (Community Health Leaders)

* Residents of the rural areas of study sites
* Voluntary participation in the monitoring of patients using the mobile app

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The effectiveness of community-based intervention using the Guaral+ST mobile application was evaluated by four outcomes: i. The number of follow-ups | 6 months
  The number of follow-up contacts between patients and health system or community health workers.
ii. Percent adherence to treatment | 6 months
  Relation between the number of doses administrated and the number of doses formulated by the physicians x 100.
iii. Adverse drug reactions | 6 months
  Frequency of adverse drug reactions: number of adverse drug reactions
iv. Therapeutic response | 6 months
  * Cure: Completely re-epithelialised lesions on days 90 -180 after initiation of treatment
  * Failure: >50% increase in ulcer size from baseline at any time during evaluation or incomplete re-epithelialised on days 90-180

SECONDARY OUTCOMES:
Implementation of the community-based strategy to follow patients with cutaneous Leishmaniasis was evaluated by three outcomes. i. Acceptability | 6 months
  It refers to the perception among implementation stakeholders that the app is appealing, suitable, or satisfactory by a qualitative evaluation at three levels: community health leaders, health workers, and, and patients.
ii. Usability | 6 months
  Refers to the degree to which the app can be used by community health leaders and health workers to achieve quantified objectives of effectiveness, efficiency, and satisfaction. It was evaluated using qualitatively at two levels: community health leaders and health workers.
iii. Fidelity | 6 months
  It refers to the compliance (percentage) with the implementation strategy as described in the protocol. It was measured at two levels: Community Health Leaders and physicians.

CONTACTS AND LOCATIONS:
Locations (1):
- Corporación Centro Internacional de entrenamiento e Investigaciónes Médicas, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navarro A, Rubiano L, Arango JD, Rojas CA, Alexander N, Saravia NG, Aronoff-Spencer E. Developing mobile health applications for neglected tropical disease research. PLoS Negl Trop Dis. 2018 Nov 1;12(11):e0006791. doi: 10.1371/journal.pntd.0006791. eCollection 2018 Nov. PMID 30383809
- [Background] Carrion C, Robles N, Sola-Morales O, Aymerich M, Ruiz Postigo JA. Mobile Health Strategies to Tackle Skin Neglected Tropical Diseases With Recommendations From Innovative Experiences: Systematic Review. JMIR Mhealth Uhealth. 2020 Dec 31;8(12):e22478. doi: 10.2196/22478. PMID 33382382
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Olliaro P, Grogl M, Boni M, Carvalho EM, Chebli H, Cisse M, Diro E, Fernandes Cota G, Erber AC, Gadisa E, Handjani F, Khamesipour A, Llanos-Cuentas A, Lopez Carvajal L, Grout L, Lmimouni BE, Mokni M, Nahzat MS, Ben Salah A, Ozbel Y, Pascale JM, Rizzo Molina N, Rode J, Romero G, Ruiz-Postigo JA, Gore Saravia N, Soto J, Uzun S, Mashayekhi V, Velez ID, Vogt F, Zerpa O, Arana B. Harmonized clinical trial methodologies for localized cutaneous leishmaniasis and potential for extensive network with capacities for clinical evaluation. PLoS Negl Trop Dis. 2018 Jan 12;12(1):e0006141. doi: 10.1371/journal.pntd.0006141. eCollection 2018 Jan. PMID 29329311
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Agarwal S, Perry HB, Long LA, Labrique AB. Evidence on feasibility and effective use of mHealth strategies by frontline health workers in developing countries: systematic review. Trop Med Int Health. 2015 Aug;20(8):1003-14. doi: 10.1111/tmi.12525. Epub 2015 May 14. PMID 25881735
- [Background] Mieras LF, Taal AT, Post EB, Ndeve AGZ, van Hees CLM. The Development of a Mobile Application to Support Peripheral Health Workers to Diagnose and Treat People with Skin Diseases in Resource-Poor Settings. Trop Med Infect Dis. 2018 Sep 15;3(3):102. doi: 10.3390/tropicalmed3030102. PMID 30274498